CLINICAL TRIAL: NCT02635282
Title: Intranasal Ketamine Versus Intranasal Midazolam Plus Fentanyl in Treating Pain Associated With Incision and Drainage of Abscesses in the Pediatric Emergency Department: A Randomized Controlled Trial
Brief Title: IN Ketamine Vs IN Midazolam and Fentanyl for Abscess I&D
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Tennessee (Other)
Responsible Party: Principal Investigator, Cynthia Copley, Principal Investigator, Pediatric Emergency Medicine Fellow, University of Tennessee
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-04113-FB
Record Dates: First submitted 2015-12-09; First posted 2015-12-18 (Estimated); Last update posted 2017-03-27 (Actual); Status verified 2017-03

CONDITIONS: Abscess; Pain
MeSH Terms: conditions — Abscess; Pain | interventions — Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IN fentanyl and midazolam (Active Comparator): group of patients who are randomized to receive intranasal fentanyl and midazolam
  Interventions: Drug: intranasal fentanyl; Drug: intranasal midazolam
- IN ketamine (Experimental): group of patients who are randomized to receive intranasal ketamine
  Interventions: Drug: intranasal ketamine

INTERVENTIONS:
Drug: intranasal ketamine
  Arms: IN ketamine
Drug: intranasal fentanyl
  Arms: IN fentanyl and midazolam
Drug: intranasal midazolam
  Other Names: Versed
  Arms: IN fentanyl and midazolam

SUMMARY:
The general objective of this study is to determine whether intranasal ketamine should be incorporated into formulary as an option to treat pain during minor procedures in the pediatric emergency department.

DETAILED DESCRIPTION:
In the pediatric emergency department, one of the main goals in patient care is to provide adequate pain management. Many patients present to the emergency department with conditions or injuries that cause acute or chronic pain. Health care providers routinely aim to treat patients' pain in a timely manner after arrival to the emergency department. A common scenario occurs when a patient presents with a condition in which treatment will require that a potentially painful or anxiety-provoking procedure will be performed in the ED, and providers also strive to treat this pain and anxiety accordingly. There are several different methods for treating pain and anxiety, including multiple types of medications, which can be given orally, intravenously, intramuscularly, or intranasally. The use of intranasal medications for the treatment of pain and anxiety has been steadily increasing over the last decade, and this has been particularly helpful in the pediatric population. There are several advantages of using intranasal medications, including rapid onset, ease of administration, and lack of need for IV access.

At this time, this pediatric emergency department uses two different medications via the intranasal route of administration: fentanyl, a synthetic opiate, and midazolam, a benzodiazepine, which are used for pain control and anxiolysis, respectively, and these two medications are frequently used together. The objective of this study is to introduce ketamine as a third medication for intranasal use and to observe its effects on pain control; this medication is currently used either intravenously or intramuscularly in the investigator's ED. Ketamine is an anesthetic that has properties of analgesia and amnesia and has a generally favorable side effect profile. This study will observe the effects of using a medication that is already widely used in the investigator's ED, but it will be used via a different route of administration, offering advantages over other options. In this study, patients will be enrolled who have been diagnosed with a soft tissue abscess that will be treated with incision and drainage in the ED. Patients in one group will be given a dose of intranasal ketamine at a predetermined dose, and measured variables will include pain score, vital signs, patient and/or parent satisfaction, adverse effects, length of stay, and need for additional doses of ketamine or additional medications. This group of patients will be compared with another group of patients who will be given intranasal fentanyl and intranasal midazolam using a randomization through the RedCap system. The investigators hypothesize that the use of intranasal ketamine in this PED for treating pain associated with the minor procedure of incision and drainage of a soft tissue abscess will provide satisfactory pain control in these patients while offering advantages over other treatment options, as compared with patients treated with the current standard intranasal medications.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of abscess with planned incision and drainage of a single abscess

Exclusion Criteria:

* Fast Track patients
* Patients who have received an opioid analgesic within the previous 4 hours of time of enrollment in study
* Patients with parent or legal guardian not present to give informed consent for enrollment in study
* Non-English speaking patients and/or parent
* Patients with a contraindication for the administration of intranasal medication (nasal trauma, aberrant nasal anatomy)
* Patients with ocular injuries
* Patients with a known allergy to ketamine, fentanyl, and/or midazolam
* Pregnant females
* Patients with history of seizure disorders

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 19 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-03-23 (Actual); Study Completion 2017-03-23 (Actual)

PRIMARY OUTCOMES:
Change in pain score measured utilizing the Faces Pain Scale-Revised | before medication administered and at 30 minutes after medication administration
  The Faces Pain Scale-Revised will be used for children ages 3-7 years
Change in pain score measured utilizing the numeric pain rating scale | before medication administered and at 30 minutes after medication administration
  The numeric pain rating scale will be used in children ages 8-17 years

SECONDARY OUTCOMES:
Vital sign measurements | before medication administered and at 15 and 30 minutes after medication administration
  Temperature, heart rate, respiratory rate, oxygen saturation, and blood pressure will be measured
Sedation score using the University of Michigan Sedation Scale | before medication administered and at 15 and 30 minutes after medication administration

CONTACTS AND LOCATIONS:
Locations (1):
- Le Bonheur Children's Hospital, Memphis, Tennessee, United States

REFERENCES:
- [Background] Bailey B, Gravel J, Daoust R. Reliability of the visual analog scale in children with acute pain in the emergency department. Pain. 2012 Apr;153(4):839-842. doi: 10.1016/j.pain.2012.01.006. Epub 2012 Feb 4. PMID 22305630
- [Result] Afridi SK, Giffin NJ, Kaube H, Goadsby PJ. A randomized controlled trial of intranasal ketamine in migraine with prolonged aura. Neurology. 2013 Feb 12;80(7):642-7. doi: 10.1212/WNL.0b013e3182824e66. Epub 2013 Jan 30. PMID 23365053
- [Result] Andolfatto G, Willman E, Joo D, Miller P, Wong WB, Koehn M, Dobson R, Angus E, Moadebi S. Intranasal ketamine for analgesia in the emergency department: a prospective observational series. Acad Emerg Med. 2013 Oct;20(10):1050-4. doi: 10.1111/acem.12229. PMID 24127709
- [Result] Del Pizzo J, Callahan JM. Intranasal medications in pediatric emergency medicine. Pediatr Emerg Care. 2014 Jul;30(7):496-501; quiz 502-4. doi: 10.1097/PEC.0000000000000171. PMID 24987995